CLINICAL TRIAL: NCT05517447
Title: An Open-label Extension Study for Participants Who Completed Study IMVT-1401-3201 or Study IMVT-1401-3202 to Assess the Efficacy and Safety of Batoclimab for the Treatment of Thyroid Eye Disease (TED)
Brief Title: Extension Study to Assess Batoclimab in Participants With Thyroid Eye Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMVT-1401-3203
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Eye Disease
Keywords: Batoclimab; Thyroid eye disease; IMVT-1401; Monoclonal antibody; Autoimmune disorders; Graves' Ophthalmopathy; Graves' Orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Observational cohort (Other): Proptosis responders in feeder studies will enter in a non-treatment observational study
  Interventions: Other: Observational cohort study
- Treatment Cohort (Experimental): Proptosis non-responders in feeder studies will be administered batoclimab of 680 milligram (mg) subcutaneous (SC) for 12 weeks followed by 340 mg SC for 12 weeks
  Interventions: Drug: Batoclimab

INTERVENTIONS:
Other: Observational cohort study — Observational cohort study
  Arms: Observational cohort
Drug: Batoclimab — Batoclimab is a fully human anti-neonatal fragment crystallizable receptor (FcRn) monoclonal antibody
  Other Names: IMVT-1401
  Arms: Treatment Cohort

SUMMARY:
This is a 2-cohort (observational and treatment cohort) extension study for participants completing feeder studies (IMVT-1401-3201 or IMVT-1401-3202). The observational cohort will assess the durability of proptosis response of feeder studies off treatment. The treatment cohort will evaluate the efficacy of batoclimab as assessed by proptosis responder rate.

ELIGIBILITY:
Inclusion criteria:

For all participants:

1. Have completed the Week 24 visit of the feeder study.

For participants assigned to the Open-label Treatment Cohort:

1. Do not require immediate surgical intervention and is not planning corrective surgery/irradiation or medical therapy for TED during the course of the study.
2. Did not permanently discontinue batoclimab

Additional inclusion criteria are defined in the protocol.

Exclusion criteria:

For all participants:

1. In the Investigator's judgement, the benefits of entry in the study do not outweigh the risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-11-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Duration of proptosis response off treatment in study eye in batoclimab responder participants in the feeder studies | Up to Week 24

SECONDARY OUTCOMES:
Percentage of proptosis responders in study eye in placebo non-responder participants in the feeder studies | At Week 24
Percentage of proptosis responders in study eye in batoclimab non-responder participants in the feeder studies | At Week 24

CONTACTS AND LOCATIONS:
Locations (55):
- United States (9):
  - Site Number - 1520, Glendora, California
  - Site Number - 1501, Aurora, Colorado
  - Site Number - 1526, Livonia, Michigan
  - Site Number - 1513, Rochester, Minnesota
  - Site Number - 1540, Las Vegas, Nevada
  - Site Number - 1508, Houston, Texas
  - Site Number - 1558, Mesquite, Texas
  - Site Number - 1511, Morgantown, West Virginia
  - Site Number - 1518, Milwaukee, Wisconsin
- Site Number - 7565, Sydney, Australia
- Belgium (4):
  - Site Number - 4671, Bruges
  - Site Number - 4672, Brussels
  - Site Number - 4673, Brussels
  - Site Number - 4670, Ghent
- Georgia (4):
  - Site Number - 3454, Tbilisi
  - Site Number - 3455, Tbilisi
  - Site Number - 3450, Tbilisi
  - Site Number - 3451, Tbilisi
- Hungary (2):
  - Site Number - 7550, Budapest
  - Site Number - 7552, Pécs
- Israel (4):
  - Site Number - 4760, Ramat Gan, Tel Aviv
  - Site Number - 4764, Afula
  - Site Number - 4761, Jerusalem
  - Site Number - 4762, Petah Tikva
- Italy (7):
  - Site Number - 6207, Catania
  - Site Number - 6204, Milan
  - Site Number - 6203, Milan
  - Site Number - 6205, Napoli
  - Site Number - 6209, Palermo
  - Site Number - 6201, Pisa
  - Site Number - 6202, Rome
- Latvia (3):
  - Site Number - 9301, Ogre
  - Site Number - 9300, Riga
  - Site Number - 9302, Ventspils
- Site Number - 7570, Christchurch, New Zealand
- Poland (4):
  - Site Number - 3107, Gliwice, Silesian Voivodeship
  - Site Number - 3101, Krakow
  - Site Number - 3104, Lublin
  - Site Number - 3105, Lublin
- Site Number - 1990, San Juan, Puerto Rico
- Slovakia (3):
  - Site Number - 9200, Bratislava
  - Site Number - 9201, Bratislava
  - Site Number - 9202, Trenčín
- Spain (5):
  - Site Number - 3602, Barcelona, Catalonia
  - Site Number - 3604, Madrid
  - Site Number - 3600, Santiago de Compostela
  - Site Number - 3606, Seville
  - Site Number - 3603, Valencia
- United Kingdom (7):
  - Site Number - 7305, Guildford
  - Site Number - 7303, London
  - Site Number - 7312, London
  - Site Number - 7313, London
  - Site Number - 7300, Manchester
  - Site Number - 7302, Newcastle upon Tyne
  - Site Number - 7308, Sheffield

IPD SHARING:
Plan to Share IPD: No